CLINICAL TRIAL: NCT05815810
Title: Novel Delivery Method of Transgender Voice Therapy Using a Mobile Application
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Ithaca College (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-12024240
Record Dates: First submitted 2023-04-03; First posted 2023-04-18 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Transitioning Voice of Transgender and Gender Diverse People
Keywords: Transgender; Voice therapy; Mobile Application

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transgender and gender diverse (TGGD) individuals using the pilot app (Experimental): The investigators will develop Attuned, an open access voice and communication modification training (VCMT) app based on standard of care. Participants will undergo VCMT via the mobile application, Attuned. Participants will include healthy transgender and gender diverse (TGGD) individuals seeking voice modification to better reflect their identity.
  Interventions: Other: Attuned: A mobile application
- Transgender and gender diverse (TGGD) individuals receiving standard voice modification (Active Comparator): VCMT via speech pathology will be compared to the efficacy of an app-based VCMT program. Participants will undergo VCMT in-person. Participants will include healthy transgender and gender diverse (TGGD) individuals seeking voice modification to better reflect their identity.
  Interventions: Other: In-Person Voice Modification Therapy

INTERVENTIONS:
Other: Attuned: A mobile application — Subjects will undergo voice and communication modification therapy via the Attuned application. This consists of an 11 week program consisting of different modules to learn how to modify voice (e.g., pitch, intonation, resonance). At the end of each module, participants will be given exercises to practice what they learned.
  Arms: Transgender and gender diverse (TGGD) individuals using the pilot app
Other: In-Person Voice Modification Therapy — Subjects will undergo standard of care in-person voice modification therapy at Ithaca College.
  Arms: Transgender and gender diverse (TGGD) individuals receiving standard voice modification

SUMMARY:
The investigators hypothesize that the mobile application they developed for transgender and gender diverse individuals (TGGD) will be equivalent or better than traditional speech therapy in improving voice quality. The investigators will measure both how the participants feel about their voices and how their voice actually sounds to see if the app is effective.

DETAILED DESCRIPTION:
The ultimate objective of this study is to use Community-Based Participatory Research (CBPR) methods to develop an effective user-friendly, health literate, inclusive and accessible mobile application (app) to improve access to gender affirming voice modification training for transgender and gender diverse (TGGD) individuals. The immediate objectives are to understand the needs of TGGD individuals in voice care,and identify barriers to creating a pilot app with evidence-based educational content for VCMT and to evaluate subjective and objective voice outcomes of TGGD participants with app use compared to standard behavioral intervention with a speech pathologist.

ELIGIBILITY:
Inclusion Criteria:

* Identify as a transgender individual
* Be 18 years or older
* Be able to read and write in English
* Have an iOS or Android Device

Exclusion Criteria:

* Identify as cisgender
* Experience hoarseness
* Experiencing any physical pain related to voice use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender and non-binary individuals
Enrollment: 50 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in Transsexual Voice Questionnaire (TVQ) Scores | Baseline, Week 4, Week 11
  The Transsexual Voice Questionnaire (TVQ) is a 30-item questionnaire that assesses self-perception of voice in transgender individuals. Responses range from (1) rarely or never to (4) usually or always. Scores range from 30 (no perceived voice difficulty) to 120 (high perceived voice difficulty).
Change in Transgender Self Evaluation Questionnaire (TSEQ) Scores | Baseline, Week 4, Week 11
  The Transgender Self Evaluation Questionnaire (TSEQ) is a 30-item questionnaire that assesses self perception in transgender and gender diverse individuals. Responses range from (1) never (4) always. Scores range from 30 (low voice satisfaction) to 120 (high voice satisfaction)
Change in Fundamental Frequency | Baseline, Week 4, Week 11
  The acoustic measure fundamental frequency will be obtained by analyzing participant's voice recordings via multi-speech acoustic analyses program of Kay-Pentax
Change in Formants | Baseline, Week 4, Week 11
  The acoustic measure formants will be obtained by analyzing participant's voice recordings via multi-speech acoustic analyses program of Kay-Pentax

SECONDARY OUTCOMES:
Usability of Mobile Application as measured by the Mobile Application Rating Scale (MARS) | Week 11
  The Mobile Application Rating Scale (MARS) is a 19-item scale that allows app users to rate the usability of a mobile application. Responses range from 1 (inadequate) to 5 (excellent). Scores range from 19-95 with a score of 19 corresponding to a poor and inadequate app and 95 of an excellent apps with great usability.

CONTACTS AND LOCATIONS:
Overall Officials: Anaïs Rameau, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Ithaca College, Ithaca, New York
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No